CLINICAL TRIAL: NCT00291525
Title: Prospective Randomized On-X Anticoagulation Clinical Trial (PROACT)
Brief Title: Randomized On-X Anticoagulation Trial
Acronym: PROACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: On-X Life Technologies, Inc. (Industry)
Collaborators: Clinipace Worldwide (Industry); Acelis Connected Health (Unknown); WCG IRB (Unknown); Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-01; G050208 (Other: FDA)
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-10

CONDITIONS: Heart Valve Disease
Keywords: valve; prosthesis; antithrombotics; randomized
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Masking Description: Number of participants below refers to randomized in all 3 study arms
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AVR Low Risk without warfarin (Experimental): AVR Low Risk without warfarin
  Interventions: Device: On-X valve using reduced anticoagulation
- AVR low risk with standard warfarin (Active Comparator): AVR low risk with standard warfarin
  Interventions: Device: On-X Valve with Standard warfarin Therapy
- AVR High risk with lower warfarin (Experimental): AVR High risk with lower warfarin
  Interventions: Device: On-X valve using reduced anticoagulation
- AVR High Risk with standard warfarin (Active Comparator): AVR High Risk with standard warfarin
  Interventions: Device: On-X Valve with Standard warfarin Therapy
- MVR with lower warfarin (Experimental): MVR with lower warfarin
  Interventions: Device: On-X valve using reduced anticoagulation
- MVR with standard warfarin (Active Comparator): MVR with standard warfarin
  Interventions: Device: On-X Valve with Standard warfarin Therapy

INTERVENTIONS:
Device: On-X valve using reduced anticoagulation — Valve replacement with antiplatelet agents or lowered warfarin
  Other Names: On-X Prosthetic Heart Valve
  Arms: AVR High risk with lower warfarin; AVR Low Risk without warfarin; MVR with lower warfarin
Device: On-X Valve with Standard warfarin Therapy — Valve replacement with standard dosage warfarin
  Other Names: On-X Prosthetic Heart Valve
  Arms: AVR High Risk with standard warfarin; AVR low risk with standard warfarin; MVR with standard warfarin

SUMMARY:
Various patient groups with the On-X Valve can be maintained safely on lower doses of blood thinner(Coumadin®) or on antiplatelet drugs (aspirin/Plavix®) only rather than the standard dose of Coumadin and aspirin presently recommended by ACC/AHA or ACCP professional societies.

DETAILED DESCRIPTION:
This is a longitudinal, randomized (randomization to occur at the 3-month follow-up) study comparing the On-X valve on low dose anticoagulation (test group) to concomitant control groups of On-X valves receiving standard Coumadin/aspirin therapy, and also to FDA objective performance criteria (OPC) for heart valve replacement. It is a multicenter study consisting of up to 50 centers in the United States, Canada, and Italy enrolling and randomizing no more than 1200 patients (200 in each of 6 groups). There are three test arms of the study: low risk aortic valve replacement, high risk aortic valve replacement, and mitral valve replacement. Each arm has an equivalent control. Test therapies are: low risk aortic valve replacement - aspirin/Plavix, high risk aortic valve replacement - Coumadin at INR of 1.5 to 2.0 plus aspirin, and mitral valve replacement - Coumadin at an INR of 2.0 to 2.5 plus aspirin. Follow-up will run for up to 8 years in each patient. Each arm is independent and the low risk aortic and high risk aortic arms are completed. The low risk aortic arm was closed early resulting in a reduction of the estimated total enrollment with randomization to 1000. The high risk arm is completed with FDA review and this arm had 375 randomized enrollees. The mitral arm continues to enroll with a planned randomized enrollment of 400.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring isolated aortic valve replacement (AVR), or isolated mitral valve replacement (MVR).
* AVR patients receiving low dose or antiplatelet only anticoagulation will be divided into groups at low risk and high risk for thromboembolism with all patients being in the low risk group except for patients with the following conditions which place a patient in the high risk group:

  * Chronic atrial fibrillation
  * Left ventricular ejection fraction < 30 %
  * Enlarged left atrium >50mm diameter
  * Spontaneous echo contrasts in the left atrium
  * Vascular pathology
  * Neurological events
  * Hypercoagulability
  * Left or right ventricular aneurysm
  * Lack of platelet response to aspirin or clopidogrel
  * Women receiving estrogen replacement therapy
* Concomitant cardiac surgery is allowed
* Adult patients

Exclusion Criteria:

* Right side valve replacement
* Double (aortic plus mitral) valve replacement
* Patients with active endocarditis at the time of implant
* Previous confirmed or suspected thromboembolic event or thrombophlebitis
* Other terminal illness
* Patients who are in an emergency state
* Inability to return for required follow-ups
* Patients with an On-X valve implanted within the study and subsequently explanted
* Patients who are known to be pregnant, plan to become pregnant or are lactating
* Patients with acquired immunodeficiency syndrome or know to be HIV positive
* Patients who are prison inmates or known drug or alcohol abusers
* Patients unable to give adequate informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2006-06-06 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Puskas, MD, Study Director — MOUNT SINAI HOSPITAL
Locations (49):
- United States (44):
  - Tucson Medical Center, Tucson, Arizona
  - Southern Arizona VA Medical Center, Tucson, Arizona
  - Loma Linda University, Loma Linda, California
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Health Care Services, Newark, Delaware
  - Medstar Heart & Vascular Institute, Washington D.C., District of Columbia
  - Shands Hospital - University of Florida, Gainesville, Florida
  - Cardiac Surgical Associates, Kissimmee, Florida
  - South Florida Heart & Lung, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - St. Francis Heart Center, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Mid America Heart institute, Kansas City, Missouri
  - Barnes Jewish Hospital - Washington University, St Louis, Missouri
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - St. Luke's Roosevelt, New York, New York
  - Montefiore Medical Center, New York, New York
  - WakeMed, Raleigh, North Carolina
  - Duke University Medical Center, Raleigh, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - University Hospital - Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma/VA Oklahoma City, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - Texas Cardiac Center, Lubbock, Texas
  - Baylor Scott & White - Plano, Plano, Texas
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - MultiCare Health System, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
  - St. Luke's Aurora Health Care, Milwaukee, Wisconsin
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - London Health Science Centre, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - IUCPQ Chirurgie Cardiaque, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puskas JD; PROACT Investigators. Reply: Low-Thrombogenicity Mechanical Heart Valves: Which Antithrombotic Strategy? J Am Coll Cardiol. 2018 Oct 9;72(15):1879-1880. doi: 10.1016/j.jacc.2018.07.063. No abstract available. PMID 30286937
- [Result] Puskas J, Gerdisch M, Nichols D, Quinn R, Anderson C, Rhenman B, Fermin L, McGrath M, Kong B, Hughes C, Sethi G, Wait M, Martin T, Graeve A; PROACT Investigators. Reduced anticoagulation after mechanical aortic valve replacement: interim results from the prospective randomized on-X valve anticoagulation clinical trial randomized Food and Drug Administration investigational device exemption trial. J Thorac Cardiovasc Surg. 2014 Apr;147(4):1202-1210; discussion 1210-1. doi: 10.1016/j.jtcvs.2014.01.004. Epub 2014 Jan 12. PMID 24512654
- [Result] Yanagawa B, Levitsky S, Puskas JD; PROACT Investigators. Reduced anticoagulation is safe in high-risk patients with the On-X mechanical aortic valve. Curr Opin Cardiol. 2015 Mar;30(2):140-145. doi: 10.1097/HCO.0000000000000149. PMID 29504958
- [Result] Puskas JD, Gerdisch M, Nichols D, Fermin L, Rhenman B, Kapoor D, Copeland J, Quinn R, Hughes GC, Azar H, McGrath M, Wait M, Kong B, Martin T, Douville EC, Meyer S, Ye J, Jamieson WRE, Landvater L, Hagberg R, Trotter T, Armitage J, Askew J, Accola K, Levy P, Duncan D, Yanagawa B, Ely J, Graeve A; PROACT Investigators. Anticoagulation and Antiplatelet Strategies After On-X Mechanical Aortic Valve Replacement. J Am Coll Cardiol. 2018 Jun 19;71(24):2717-2726. doi: 10.1016/j.jacc.2018.03.535. PMID 29903344
- [Derived] Chu MWA, Ruel M, Graeve A, Gerdisch MW, Damiano RJ Jr, Smith RL 2nd, Keeling WB, Wait MA, Hagberg RC, Quinn RD, Sethi GK, Floridia R, Barreiro CJ, Pruitt AL, Accola KD, Dagenais F, Markowitz AH, Ye J, Sekela ME, Tsuda RY, Duncan DA, Swistel DG, Harville LE 3rd, DeRose JJ, Lehr EJ, Alexander JH, Puskas JD; PROACT Mitral Investigators. Low-Dose vs Standard Warfarin After Mechanical Mitral Valve Replacement: A Randomized Trial. Ann Thorac Surg. 2023 Apr;115(4):929-938. doi: 10.1016/j.athoracsur.2022.12.031. Epub 2023 Jan 4. PMID 36610532
- [Derived] Chu MWA, Ruel M, Graeve A, Gerdisch MW, Damiano RJ Jr, Smith RL 2nd, Keeling WB, Wait MA, Hagberg RC, Quinn RD, Sethi GK, Floridia R, Barreiro CJ, Pruitt AL, Accola KD, Dagenais F, Markowitz AH, Ye J, Sekela ME, Tsuda RY, Duncan DA, Swistel DG, Harville LE 3rd, DeRose JJ, Lehr EJ, Puskas JD; PROACT Mitral Investigators. WITHDRAWN: Low-Dose Versus Standard Warfarin After Mechanical Mitral Valve Replacement: A Randomized Controlled Trial. Ann Thorac Surg. 2022 Jan 28:S0003-4975(22)00138-2. doi: 10.1016/j.athoracsur.2022.01.015. Online ahead of print. PMID 35101419

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
Started | 99 | 102 | 185 | 190 | 201 | 200
Completed | 19 | 74 | 81 | 112 | 132 | 120
Not Completed | 80 | 28 | 104 | 78 | 69 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin | Total
Number analyzed (Participants) | 99 | 102 | 185 | 190 | 201 | 200 | 977
Age, Customized [Mean (Standard Deviation); unit: years] | 53.5 (10.9) | 52.5 (11.6) | 54.1 (13.0) | 55.8 (12.0) | 55.0 (11.2) | 54.9 (11.6) | 54.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 37 | 36 | 121 | 124 | 367
  Male | 76 | 76 | 148 | 154 | 80 | 76 | 610
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Thromboembolism
Description: Percentage of events per patient year
Time Frame: 8 years
Measure: Number; unit: %/patient years
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
Number analyzed (Participants) | 99 | 102 | 185 | 190 | 201 | 200
%/patient years | 4.86 | 0.29 | 2.43 | 1.74 | 2.48 | 2.08

2. Primary Outcome: Valve Thrombosis
Description: Percentage of events per patient year
Time Frame: 8 years
Population: Numbers in parentheses are Linearized Occurrence Rates (LOR)
Measure: Number; unit: %/patient years
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
Number analyzed (Participants) | 99 | 102 | 185 | 190 | 201 | 200
%/patient years | 0.69 | 0.87 | 0.21 | 0.37 | 0.46 | 0.40

3. Primary Outcome: Bleeding Events
Description: Percentage of events per patient year
Time Frame: 8 years
Measure: Number; unit: Linearized Occurrence Rates (LOR): %/pat
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
Number analyzed (Participants) | 99 | 102 | 185 | 190 | 201 | 200
Linearized Occurrence Rates (LOR): %/pat | 3.82 | 3.49 | 2.86 | 7.43 | 9.63 | 10.01

4. Secondary Outcome: Valve-Related Mortality
Description: Percentage of events per patient year
Time Frame: 8 years
Measure: Number; unit: %/patient years
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
Number analyzed (Participants) | 99 | 102 | 185 | 190 | 201 | 200
%/patient years | 0.69 | 0.87 | 0.21 | 0.37 | 0.28 | 0.10

5. Secondary Outcome: Valve Hemodynamics
Description: Echocardiograpic measures of valve hemodynamics at 5 years
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
Number analyzed (Participants) | 99 | 102 | 185 | 190 | 201 | 200
mmHg
  Peak Gradient mmHg | 22.64 (11.74) | 21.31 (12.24) | 15.8 (9.8) | 16.7 (8.5) | 11.9 (4.4) | 12.6 (7.5)
  Mean Gradient mmHg | 11.38 (6.25) | 11.00 (5.87) | 7.6 (5.0) | 8.8 (4.2) | 4.6 (1.93) | 4.7 (1.98)

ADVERSE EVENTS:
Time Frame: Events occurrence rate is presented for each arm at the end of its follow-up period. Time frame/Follow-up duration is different for each study arms (due to dependency on enrollment rate and timing of follow-up cessation at each arm): Aortic arm Low Risk: 8.6 years Aortic arm High Risk: 9.2 years Mitral arm: 14.7
Description: Adverse events are reported as simple occurrence rates.
  "Other" Adverse Events were not collected in this study; only risks/events that are known as associated with heart valve replacement were reported and adjudicated (presented above). Classification of events was based on the AATS/STS guidelines categories and definitions rather than on serious/non-serious. The number of "Other" AEs is reported here as "0" because none were collected in the study.
Arm/Group | AVR Low Risk Without Warfarin | AVR Low Risk With Standard Warfarin | AVR High Risk With Lower Warfarin | AVR High Risk With Standard Warfarin | MVR With Lower Warfarin | MVR With Standard Warfarin
All-Cause Mortality (participants affected / at risk) | 5/99 | 4/102 | 10/185 | 9/190 | 17/201 | 23/200
Serious Adverse Events (participants affected / at risk) | 13/99 | 13/102 | 38/185 | 43/190 | 94/201 | 89/200
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVR Low Risk Without Warfarin (N=99) | AVR Low Risk With Standard Warfarin (N=102) | AVR High Risk With Lower Warfarin (N=185) | AVR High Risk With Standard Warfarin (N=190) | MVR With Lower Warfarin (N=201) | MVR With Standard Warfarin (N=200)
Paravaluvular Leak (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 5 (5) | 1 (1) — "Any evidence of leakage of blood around the prosthesis between the sewing ring and native annulus" (Protocol, Section C, page 21
Endocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 10 (10) — Documented evidence of infection of the prosthesis [Protocol, Section C, page 20]
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 10 (10) | 31 (31) | 33 (33) — Whether considered valve-related or not
Other - Cardiovascular and Pulmonary (Cardiac disorders) | 10 (10) | 12 (12) | 27 (27) | 25 (25) | 55 (55) | 45 (45) — Complication or any new diagnosis that is not related to the prosthesis, but is important to subsequent morbidity and mortality of the patient (Protocol, Section C, Page 22)

LIMITATIONS AND CAVEATS:
1. Study collected/reported events based on AATS/STS Guidelines (events of interest, with no serious/non-serious distinction).
2. Enrollment started 2006 for 3 arms:

   AVR Low Risk - Enrollment & follow-up terminated 2014, indication not pursued AVR High Risk - Enrollment ended 2009, follow up completed 2014, low INR indication granted MVR - Enrollment ended 2020, follow up completed 2023, indication not pursued
3. Total SAEs is total of all categories presented minus mortality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-03-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT00291525/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2011-04-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT00291525/SAP_001.pdf